CLINICAL TRIAL: NCT02150486
Title: Postoperative Myocardial Injury and Non-cardiac Complications After Major Abdominal Surgery in Patients at Risk for Coronary Artery Disease
Brief Title: Myocardial Injury and Postoperative Complications
Acronym: MICOLON
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, MD PhD, St. Antonius Hospital
Other Study IDs: NL39172.100.11
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether perioperative myocardial injury is associated with adverse outcome in patients scheduled for major abdominal surgery.

DETAILED DESCRIPTION:
Study design

The MICOLON study is a prospective, single-centre, observational cohort study on the association between 5th generation high sensitive cardiac troponin T levels and non-cardiac outcome after major abdominal surgery in patients at risk for coronary artery disease.

Patient eligibility

Patients are eligible to enter the study if they are scheduled to undergo elective major abdominal surgery with an expected postoperative mortality rate >3%, are aged 45 years or older and have at least one of the following major cardiac risk factors: diabetes mellitus, peripheral artery disease (i.e. intermittent claudication or history of vascular surgery except arteriovenous shunt and vein stripping procedures), history of hospitalization for congestive heart failure, history of myocardial infarction, stable angina pectoris, history of coronary artery bypass grafting or percutaneous coronary angioplasty, renal insufficiency (defined as preoperative creatinine >150 μmol/L), history of cerebral vascular event, aortic valve stenosis (defined as aortic valve area <1 cm2), atrial fibrillation, moderate or poor left ventricular function (defined as left ventricular ejection fraction <55%), or two of the following minor risk factors for coronary artery disease: age >70 years, hypertension, hypercholesterolemia, history of transient ischemic attack, chronic obstructive pulmonary disease, smoking or low functional capacity (capable of physical activity of 4 metabolic equivalents or less). Patients are excluded from study participation if they have no signed informed consent.

Study procedure

Patients eligible for the study are identified at the outpatient preoperative anesthesiology clinic. Patients are examined and screened for cardiac risk factors by an anesthesiology resident or a dedicated screening nurse. Results of preoperative laboratory tests, data on patient characteristics and preoperative use of cardiovascular drugs (i.e. statin, ß--blocker, platelet inhibitor, calcium antagonists, angiotensin-converting enzyme inhibitor and angiotensine receptor blocker) were noted. Prior to any study procedure written informed consent is obtained from all patients. During the study period blood is collected for plasma troponin T measurements after induction of general anesthesia (baseline) and on the 1st, 3rd and 7th postoperative day. All plasma samples are frozen and stored at -20°C at the hospital's laboratory until analysis. Cardiac troponin T batch analysis is performed every 3 weeks with the use of 5th generation Elecsys Troponin T high sensitive assay on an automated Cobas 6000 platform (Roche Diagnostics, Germany). The limit of detection of this high sensitive assay was determined at 3 ng/L with a 99th percentile upper reference limit of 14 ng/L. In addition, plasma creatinine levels are measured in each sample with an enzymatic method on the same automated platform (Roche Diagnostics, Germany). An estimated glomerular filtration rate is calculated from plasma creatinine values using the Modification of Diet in Renal Disease formula. During the entire study period daily routine quality control samples for troponin and creatinine ensure comparable patient data across different reagent lots. After analysis the samples are stored at -80°C.

Surgical procedures are performed under general anesthesia or a combination of general and epidural anesthesia. Anesthesia management is left to the discretion of the attending anesthesiologist. According to hospital protocol, patients scheduled for gastric-esophageal, pancreatic or hepatic surgery and patients aged ≥80 or with an American Association of Anesthesiologists physical status classification system ≥3 will be admitted to an intensive care unit postoperatively for at least 24 hours. To improve postoperative recovery all patients are treated according to the current Enhanced Recovery After Surgery guidelines.

During the postoperative period research personnel performs patient visits, reviews medical charts and notes complications. At thirty days after surgery troponin results are reported to the researchers and a follow-up telephone interview is performed if patients are discharged from the hospital at that time. Patients will be asked if a medical complication has occurred since their discharge from the hospital. If so, medical details are retrieved from their treating physicians. Information from routine postoperative clinic visits is used if patients can not be reached by telephone. Noted endpoints are judged by an event committee, that is blinded for troponin results.

Endpoint definition

Primary parameter of the study is postoperative myocardial injury at day 1, 3 or 7. Secondary parameters are met by the occurrence of any of the following non-cardiac events within 30 days after surgery: mortality - defined as death without cardiovascular origin; sepsis - defined as systemic inflammatory response syndrome (SIRS) in response to a proven or suspected microbial infection; pneumonia - defined as purulent sputum or isolation of a pathogen from sputum culture or blood culture and clinical symptoms (e.g. dyspnea, fever, cough) or a consolidation or pleural effusion on chest radiograph; respiratory failure - defined as non-cardiac hypoxia or hypercapnia leading to ICU (re)admission for respiratory support (e.g. (non)invasive ventilation or high concentration oxygen therapy); anastomotic dehiscence - defined as presence of luminal contents through drain or wound site causing local inflammation or SIRS, or leak detected on imaging studies in combination with clinical signs of SIRS; intestinal ischemia - defined as signs of superficial or transmural bowel ischemia on imaging studies and clinical symptoms (e.g. abdominal pain or tenderness) or SIRS; wound infection - purulent drainage from superficial incision or deliberate opening of superficial incision by surgeon and clinical signs of local inflammation (e.g. pain, tenderness, swelling, redness); bleeding - defined as abnormal postoperative bleeding needing surgical (i.e. re-operation) or endovascular (i.e. coiling) treatment. Other study parameters were length of hospital stay and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 45 years of age with 1 or more major cardiovascular risk factors: Congestive heart failure, peripheral artery disease (intermittent claudication, history of vascular surgery etc), diabetes mellitus type I or II, coronary artery disease (history of myocardial infarction, stable angina pectoris, history of ischemia or coronary artery disease on cardiac tests (electrocardiogram, scintigraphy, echocardiogram, coronary angiogram etc), cerebrovascular accident, renal insufficiency (creatinine > 150umol/l), aortic valve stenosis (valve area < 1 cm2) OR 2 or more minor cardiovascular risk factors: Age > 70, hypertension, high cholesterol, low functional capacity (4 metabolic equivalents or less), transient ischemic attack, chronic obstructive pulmonary disease AND undergoing abdominal surgery with an expected 30-day mortality rate > 2-3%: colorectal, gastric, pancreatic and liver surgery.

Exclusion Criteria:

* Age < 45 years of age, not scheduled for higher risk abdominal surgery, low cardiovascular risk profile.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective abdominal surgery at risk for coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Postoperative myocardial injury | 7 days
  high sensitive troponin elevation at day 1, 3 or 7 after surgery

SECONDARY OUTCOMES:
Complication | 30-days
  wound infection, pneumonia, anastomotic dehiscence, sepsis, respiratory insufficiency, bleeding, intestinal ischemia, death.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Noordzij, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Derived] Noordzij PG, van Geffen O, Dijkstra IM, Boerma D, Meinders AJ, Rettig TC, Eefting FD, van Loon D, van de Garde EM, van Dongen EP. High-sensitive cardiac troponin T measurements in prediction of non-cardiac complications after major abdominal surgery. Br J Anaesth. 2015 Jun;114(6):909-18. doi: 10.1093/bja/aev027. Epub 2015 Mar 3. PMID 25740400